CLINICAL TRIAL: NCT04356313
Title: Seguridad y Eficacia de la Plataforma Gore® Excluder® Iliac Branch y análisis de su Comportamiento en Combina-ción Con la Endoprótesis GORE® VIABAHN® VBX Ba-lloon Expandable
Brief Title: Safety and Efficacy of the Gore® Excluder® Iliac Branch Platform and Analysis of Its Behavior in Combination With the GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis (IBERVIX)
Acronym: IBERVIX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asociacion para el Estudio de la Enfermedades Vasculares de Galicia (Other)
Collaborators: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: AEEVGalicia
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Aortic Aneurysm; Iliac Aneurysm
Keywords: Iliac branch device; Aoto-iliac aneurysm; Hipogastric artery
MeSH Terms: conditions — Aortic Aneurysm; Iliac Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- GORE® EXCLUDER® Iliac Branch Endoprosthesis & HGB: Patients with Aorto-Iliac Aneurysm with implantation of a Iliac Branch device (IBE) and the Hipogastric component (HGB)
  Interventions: Device: GORE® EXCLUDER® Iliac Branch Endoprosthesis
- GORE® EXCLUDER® Iliac Branch Endoprosthesis & VBx: Patients with Aorto-Iliac Aneurysm with implantation of a Iliac Branch device (IBE) and Viabahn Balloon Expandable ( VBx)
  Interventions: Device: GORE® EXCLUDER® Iliac Branch Endoprosthesis

INTERVENTIONS:
Device: GORE® EXCLUDER® Iliac Branch Endoprosthesis — Compare between patients where Gore Excluder Iliac Branch Endoprosthesis and the Hipogastric component can be used with the group where the Hipogastric component can't be used for anatomical issues and a Gore Viabahn VBX is used instead of the Hipogastric component
  Other Names: GORE® VIABAHN® VBX Balloon Expandable Endoprosthesi

SUMMARY:
Aorto-iliac aneurysms with involvement of the iliac bifurcation or hypogastric artery aneurysms constitute only 20% of all aneurysmal pathology of the abdominal aorta. As it is a rare pathology, in order to carry out a comprehensive study of the results, it is necessary to carry out multicenter studies to collect a considerable number of cases.

One of the most widely used devices worldwide is the GORE® EXCLUDER® Iliac Branch Endoprosthesis, CE marked since 2013, this stent consists of two components: the iliac branch stent and the hypogastric component (HGB), for its joint use there are instructions for use in relation to the anatomical characteristics of the patient in order to be used.

Currently, there are other devices that can be used as a hypogastric component when the patient's anatomy does not allow the use of HGB, one of them is: GORE® VIABAHN® VBX Balloon Expandable Endoprosthesis, CE marked since 2017.

This study is designed to evaluate the efficacy and safety of devices with iliac branches for the treatment of aorto-iliac aneurysms that affect the bifurcation of common iliacs, with the use of these devices, as well as to determine the quality of life of patients after their implantation.

DETAILED DESCRIPTION:
This is a multicenter study in which 10 to 15 hospitals will participate. It is a non-intervention study in which the data from the medical records of the patients will be collected according to the action protocols of each center.

This is a prospective, non-randomized study where the data of the implants performed during a 12-month period will be recorded. Both the diagnosis and the follow-up of the patients to whom the device is implanted will strictly adhere to the protocols present in each center and which are the ones used according to all current clinical guidelines. At no time will any intervention or diagnostic test be performed outside the protocols in force in each center. The study does not imply any intervention or visit for the participants that is not routine clinical practice according to the clinical-healthcare procedures of each participating center.

Following routine clinical evaluations performed as part of standard patient care, it will be decided, after obtaining informed consent from patients, and whether they are eligible for the study and scheduled for the implant procedure with the devices. of the study.

After a baseline evaluation, the implant will be performed according to the usual clinical practice of each participating center. A follow-up visit will be made 30 days, 6 and 12 months after the procedure.

Investigators will perform implant and device evaluations and document adverse events (AE) and possible device deficiencies

Study objectives

1. Primary Objectives 1.1. General safety and efficacy at 6 months post-implant

Defined as :

* Absence of symptoms or rupture of the aneurysm.
* Growth of the aneurysm.
* Absence of reintervention.
* Need for conversion to open surgery.
* Significant clinical migration.
* Branch occlusions.

1.2 Technical success: GORE® Excluder® IBE implant in the planned location. No conversion, death, type I or III endoleaks or obstruction of the extremity of the graft.

1.3. Safety and efficacy of IBE together with VBX compared to IBE all-in-one system at 6 months.

2 Secondary objectives 2.1. Absence of major adverse effects defined as:

* Absence of morbidity and / or mortality related to the aneurysm or the device.
* Absence of mortality from any cause.

2.2. Assessment of quality of life based on the EuroQol 5D questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Patients who have an aortoiliac aneurysm with criteria to be operated electively and who meet the anatomical criteria to be treated with the devices under study within the instructions for use.

Exclusion Criteria:

* Patients who, given their anatomical characteristics, do not comply with the instructions for use of the devices under study.
* Patients with pathology at the iliac level but not aneurysmal.
* Patients who do not sign the informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have an aortoiliac aneurysm with criteria to be operated electively and who meet the anatomical criteria to be treated with the devices under study within the instructions for use treated in the participants Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
General safety and efficacy at 6 months post-implant | 6 months
  Absence of symptoms or rupture of the aneurysm. Growth of the aneurysm. Absence of reintervention. Need for conversion to open surgery. Significant clinical migration. Branch occlusions
Technical success | 1 year
  GORE® Excluder® IBE implant in the planned location. No conversion, death, type I or III endoleaks or obstruction of the extremity of the graft.
Safety and efficacy | 6 months
  IBE together with VBX compared to IBE all-in-one system

SECONDARY OUTCOMES:
Absence of major adverse effects | 6 months
  Absence of morbidity and / or mortality related to the aneurysm or the device. Absence of mortality from any cause.
Assessment of quality of life | 6 months
  Based on the EuroQol 5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Fernández Noya, M.D, Principal Investigator — University Clinical Hospital- Santiago de Compostela
Locations (1):
- University Clinical Hospital, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided